CLINICAL TRIAL: NCT04454138
Title: Ab Interno Gelatin Stent With Mitomycin C Using Targeted Supra-tenon's Placement
Status: Completed | Type: Observational
Sponsor: Prism Eye Institute (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Iqbal Ahmed, Principal Investigator, Prism Eye Institute
Other Study IDs: 955
Record Dates: First submitted 2020-06-23; First posted 2020-07-01 (Actual); Results first posted 2020-08-05 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Targeted supratenon's placement of XEN 45: Placement of Xen-45 gelatin microstent in the supra-tenon's space to maximize aqueous outflow, while preventing obstruction, limiting fibrosis of the bleb, and promoting long-term patency.
  Interventions: Device: XEN-45 gelatin microstent
- Non-targeted placement of XEN 45: Implantation of the XEN-45 gelatin microstent within the subconjunctival space, avoiding intra-tenon's placement.
  Interventions: Device: XEN-45 gelatin microstent

INTERVENTIONS:
Device: XEN-45 gelatin microstent — Placement either in the subconjunctival space or supratenon's area

SUMMARY:
The Xen-45 gelatin microstent is a novel, bleb-forming microinvasive glaucoma surgery (MIGS). Despite demonstrating similar efficacy and safety to trabeculectomy (traditional surgery), the Xen-45 gelatin microstent continues to suffer from occasional surgical failure due to fibrosis of the filtering bleb, and obstruction of the stent. During surgery, placement in a surgery known as supra-tenon's space is believed to maximize aqueous outflow, while preventing obstruction, limiting fibrosis of the bleb, and promoting long-term patency. Despite the theoretical merits, long-term data of outcomes after targeted supra-tenon's placement is needed to fully assess its potential in improving Xen-45 microstent outcomes.

DETAILED DESCRIPTION:
The Xen-45 gelatin microstent (Allergan, Dublin, Ireland) is a novel, bleb-forming microinvasive glaucoma surgery (MIGS). Creation of a filtering bleb through the gel stent and under the conjunctiva lowers intraocular pressure (IOP) by bypassing the natural outflow pathway of aqueous. A recent retrospective cohort study showed comparable safety and risk of failure to trabeculectomy. Amongst the main advantages of this device is the ability to create a bleb without dissecting and disrupting tissue, thus decreasing the amount of wound healing and potentially limiting bleb failure. However, despite demonstrating similar efficacy and safety to trabeculectomy,2 the Xen-45 gelatin microstent continues to suffer from occasional surgical failure due to fibrosis of the filtering bleb, and obstruction of the stent. Although antimetabolites, such as mitomycin C, have decreased reactionary wound healing that can result following surgery, fibrosis may still occur, especially when the components of the Xen-45 gelatin microstent are in close proximity to the fibroblastic structures of tenon's fascia.Tenon's capsule resembles a sponge-like layer with multiple adhesions to the overlying conjunctiva and underlying episclera. Implantation of the XEN within this space creates a higher risk of obstruction and subsequent failure. To ensure the lowest potential for occlusion, bleb scarring, and failure, one must ensure careful placement of the device in the subconjunctival space, avoiding intra-tenon's placement. Placement in the supra-tenon's space is believed to maximize aqueous outflow, while preventing obstruction, limiting fibrosis of the bleb, and promoting long-term patency. Despite the theoretical merits, long-term data of outcomes after targeted supra-tenon's placement is needed to fully assess its potential in improving Xen-45 microstent outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 30-90 with primary or pigmentary/pseudoexfolliative open angle, primary closed angle, or combined mechanism glaucoma with IOP of 18-40 mmHg on maximum tolerated medical therapy who received a gelatin stent with MMC at Prism Eye Institute from June 2012 to August 2019.

Exclusion Criteria:

* Other forms of glaucoma
* Prior incisional glaucoma surgery
* CPC
* Prior corneal graft (PKP, DALK, DSAEK, DMEK).

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 30-90 with primary or pigmentary/pseudoexfolliative open angle, primary closed angle, or combined mechanism glaucoma with IOP of 18-40 mmHg on maximum tolerated medical therapy who received a gelatin stent with MMC at Prism Eye Institute from June 2012 to August 2019.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iqbal Ike Ahmed, MD, Principal Investigator — Prism Eye Institute
Locations (1):
- Prism Eye Institute, Oakville, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conlon R, Saheb H, Ahmed II. Glaucoma treatment trends: a review. Can J Ophthalmol. 2017 Feb;52(1):114-124. doi: 10.1016/j.jcjo.2016.07.013. Epub 2016 Nov 17. PMID 28237137
- [Background] Schlenker MB, Gulamhusein H, Conrad-Hengerer I, Somers A, Lenzhofer M, Stalmans I, Reitsamer H, Hengerer FH, Ahmed IIK. Efficacy, Safety, and Risk Factors for Failure of Standalone Ab Interno Gelatin Microstent Implantation versus Standalone Trabeculectomy. Ophthalmology. 2017 Nov;124(11):1579-1588. doi: 10.1016/j.ophtha.2017.05.004. Epub 2017 Jun 7. PMID 28601250
- [Background] Fea AM, Spinetta R, Cannizzo PML, Consolandi G, Lavia C, Aragno V, Germinetti F, Rolle T. Evaluation of Bleb Morphology and Reduction in IOP and Glaucoma Medication following Implantation of a Novel Gel Stent. J Ophthalmol. 2017;2017:9364910. doi: 10.1155/2017/9364910. Epub 2017 Jun 20. PMID 28751986
- [Background] Sng CC, Wang J, Hau S, Htoon HM, Barton K. XEN-45 collagen implant for the treatment of uveitic glaucoma. Clin Exp Ophthalmol. 2018 May;46(4):339-345. doi: 10.1111/ceo.13087. Epub 2017 Nov 29. PMID 29053204

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-targeted Placement of XEN 45 | Targeted Supratenon's Placement of XEN 45
Started | 65 | 77
Completed | 65 | 77
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-targeted Placement of XEN 45 | Targeted Supratenon's Placement of XEN 45 | Total
Number analyzed (Participants) | 65 | 77 | 142
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65.4 [55.8 to 71.6] | 78 [70 to 83.6] | 70.9 [55.8 to 83.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 36 | 63
  Male | 38 | 41 | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 11 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 2 | 10
  White | 41 | 59 | 100
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  Canada | 65 | 77 | 142
Diabetic [Count of Participants; unit: Participants] | 22 | 11 | 33
Preoperative Best Corrected Visual Acuity (BCVA) [Median (Inter-Quartile Range); unit: logMAR] | 0.2 [0.1 to 0.3] | 0.3 [0.2 to 0.5] | 0.2 [0.0 to 0.5]
Number of Patients who received XEN 45 in Left Eye [Count of Participants; unit: Participants] | 32 | 36 | 68
IOP > 21 mmHg [Count of Participants; unit: Participants] | 32 | 42 | 74
IOP median [Median (Inter-Quartile Range); unit: mmHg] | 21 [18 to 27.5] | 22 [19.5 to 26] | 21 [18 to 27.5]
Medication Classes [Median (Inter-Quartile Range); unit: Medication Classes] | 4 [3 to 4] | 4 [2 to 4] | 4 [2 to 4]
Primary Open Angle Glaucoma [Count of Participants; unit: Participants] | 48 | 42 | 90
Pseudoexfoliation [Count of Participants; unit: Participants] | 7 | 21 | 28
Pigment Dispersion Glaucoma [Count of Participants; unit: Participants] | 3 | 0 | 3
Primary Angle Closure Glaucoma [Count of Participants; unit: Participants] | 1 | 7 | 8
Combined Mechanism Glaucoma [Count of Participants; unit: Participants] | 6 | 7 | 13
Cup to Disk Ratio [Median (Inter-Quartile Range); unit: Ratio] | 0.9 [0.8 to 0.9] | 0.8 [0.7 to 0.9] | 0.8 [0.7 to 0.9]
Preoperative Mean Deviation on Visual Field to Normal Population [Median (Inter-Quartile Range); unit: decibel] | -8.4 [-14.1 to -4.2] | -1.7 [-8 to 0] | -4 [-14.1 to 0]
Mild Disease [Count of Participants; unit: Participants] — 0 to >-6.0 dB mean deviation from normal in visual fields
  Participants | 22 | 52 | 74
Moderate to Severe Disease [Count of Participants; unit: Participants] — ≤-6.0 dB mean deviation from normal visual fields
  Participants | 42 | 25 | 67
Laser Peripheral Iridotomy [Count of Participants; unit: Participants] | 8 | 16 | 24
Laser Trabeculoplasty [Count of Participants; unit: Participants] | 47 | 41 | 88
Concomitant Cataract Surgery [Count of Participants; unit: Participants] | 24 | 38 | 62

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Intraocular Pressure Changes Between Targeted Supratenon's Placement of XEN-45 Gelatin Stent and Nontargeted Placement.
Description: Mean change in IOP from baseline, IOP thresholds of ≥6 and ≤14 (mmHg) on no medications
Time Frame: Post op year 1
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Non-targeted Placement of XEN 45 | Targeted Supratenon's Placement of XEN 45
Number analyzed (Participants) | 65 | 77
Participants | 20 | 15

2. Primary Outcome: Postoperative Intraocular Pressure Changes Between Targeted Supratenon's Placement of XEN-45 Gelatin Stent and Nontargeted Placement 2.
Description: Mean change in IOP from baseline, IOP thresholds of ≥6 and ≤14 (mmHg) +/- Medications
Time Frame: Post op Year 1
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Non-targeted Placement of XEN 45 | Targeted Supratenon's Placement of XEN 45
Number analyzed (Participants) | 65 | 77
Participants | 33 | 22

3. Primary Outcome: Postoperative Intraocular Pressure Changes Between Targeted Supratenon's Placement of XEN-45 Gelatin Stent and Nontargeted Placement 3.
Description: Mean change in IOP from baseline, IOP thresholds of ≥6 and ≤17 (mmHg) on no medications
Time Frame: Post op year 1
Population: Per protocol polulation
Measure: Count of Participants; unit: Participants
Arm/Group | Non-targeted Placement of XEN 45 | Targeted Supratenon's Placement of XEN 45
Number analyzed (Participants) | 65 | 77
Participants | 28 | 18

4. Primary Outcome: Postoperative Intraocular Pressure Changes Between Targeted Supratenon's Placement of XEN-45 Gelatin Stent and Nontargeted Placement 4.
Description: Mean change in IOP from baseline, IOP thresholds of ≥6 and ≤17 (mmHg) +/- medication
Time Frame: Post op Year 1
Population: per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Non-targeted Placement of XEN 45 | Targeted Supratenon's Placement of XEN 45
Number analyzed (Participants) | 65 | 77
Participants | 41 | 26

5. Primary Outcome: Postoperative Intraocular Pressure Changes Between Targeted Supratenon's Placement of XEN-45 Gelatin Stent and Nontargeted Placement 5.
Description: Mean change in IOP from baseline, IOP thresholds of ≥6 and ≤21 (mmHg) on no medications
Time Frame: Post op Year 1
Population: per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Non-targeted Placement of XEN 45 | Targeted Supratenon's Placement of XEN 45
Number analyzed (Participants) | 65 | 77
Participants | 31 | 19

6. Primary Outcome: Postoperative Intraocular Pressure Changes Between Targeted Supratenon's Placement of XEN-45 Gelatin Stent and Nontargeted Placement 6.
Description: Mean change in IOP from baseline, IOP thresholds of ≥6 and ≤14 (mmHg) +/- medications
Time Frame: Post op year 1
Population: per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Non-targeted Placement of XEN 45 | Targeted Supratenon's Placement of XEN 45
Number analyzed (Participants) | 65 | 77
Participants | 47 | 28

7. Secondary Outcome: Number of Participants With Postoperative Complications Between Targeted Supratenon's Placement of XEN-45 Gelatin Stent and Non-targeted Placement.
Description: Presence or absence of the following complications:
  i. Starting after POM1: shallow AC w/ iridocorneal touch, any hyphema, corneal edema, wound leak/dehiscience, choroidal effusion, malignant glaucoma, dellen/non-healing epithelial defect, ptosis, diplopia.
  ii. At any point: additional glaucoma surgery, loss of light perception vision, vitreous hemorrhage, ≥2mm hyphema, hypotony maculopathy, implant migration/blockage/exposure/extrusion, macular edema, choroidal effusion/hemorrhage requiring drainage, suprachoroidal hemorrhage, retinal detachment, suture abscess/blebitis/endophthalmitis
Time Frame: Post op year 1
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Non-targeted Placement of XEN 45 | Targeted Supratenon's Placement of XEN 45
Number analyzed (Participants) | 65 | 77
Participants | 35 | 48

8. Secondary Outcome: Number of Participants With Postoperative Interventions Between Targeted Supratenon's Placement of XEN-45 Gelatin Stent and Non-targeted Placement.
Description: Presence or absence of the following management interventions (not considered complications): bleb needling, AC reformation, suture release, digital ocular compression, use of glaucoma medications, or laser/tpa to blocked ostomy or lumen.
Time Frame: Post op year 1
Population: per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Non-targeted Placement of XEN 45 | Targeted Supratenon's Placement of XEN 45
Number analyzed (Participants) | 65 | 77
Participants | 32 | 40

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Non-targeted Placement of XEN 45 | Targeted Supratenon's Placement of XEN 45
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/77
Other Adverse Events (participants affected / at risk) | 0/65 | 0/77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/38/NCT04454138/Prot_SAP_000.pdf